CLINICAL TRIAL: NCT04134078
Title: Improving Outcomes in Cardiac Arrest With Inhaled Nitric Oxide
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Jignesh Patel, Associate Professor of Medicine, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 648019
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- inhaled nitric oxide (Experimental): Inhaled Nitric Oxide at 40 ppm will be administered in adults who suffer in hospital cardiac arrest. The administration of inhaled nitric oxide at 40 ppm will be provided upto 24 hours once ROSC is achieved.
  Interventions: Drug: inhaled nitric oxide

INTERVENTIONS:
Drug: inhaled nitric oxide — Inhaled nitric oxide at 40 ppm will be administered upto 24 hours post ROSC in patient who developed in hospital cardiac arrest

SUMMARY:
Sudden cardiac arrest (CA) is a leading cause of death worldwide. CA claims the lives of an estimated 300,000 Americans each year. Despite advances in cardiopulmonary resuscitation (CPR) methods, only approximately 10% of adults with CA survive to hospital discharge, and up to 60% of survivors have moderate to severe cognitive deficits 3 months after resuscitation. Most of the immediate and post-CA mortality and morbidity are caused by global ischemic brain injury. The goal of this grant application is to test the hypothesis that resuscitation from cardiac arrest can be improved by improving cerebral oxygenation through inhalation of nitric oxide. This strategy will also improve the chances of return of spontaneous circulation (ROSC), improve short-term survival and neurologic outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and above
2. In-hospital cardiac arrest as defined by cessation of heartbeat
3. Presence of Endotracheal Tube

Exclusion Criteria:

1. Age below 18 years
2. Absence of Endotracheal Tube
3. Patients with out-of-hospital cardiac arrest
4. Patients involved in trauma and/or patients in the SICU or CTICU
5. Preexisting intra-cerebral lesions such as any head injury (old or new), brain hematoma, cerebral hemorrhage or known frontal lobe disorders such as tumors
6. Any patient with a terminal condition that cannot be treated (specifically any terminal malignancy, end stage lung fibrosis, chronic heart failure with an ejection fraction <20%)
7. Patients with do not resuscitate and/or do not intubate (DNR/DNI) status
8. Therapeutic window has passed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Rate of return of spontanueous circulation (ROSC) | 1 day
  The primary outcome measure is to evaluate rates of return of spontaneous circulation (ROSC) from in hospital cardiac arrest patient who receive inhaled nitric oxide
Change in cerebral oxygenation (rSO2) | 1 day
  The outcomes measure is to evaluate change in the concentration of cerebral oxygenation measured by Near-infrared spectroscopy before and after the administration of inhaled nitric oxide

SECONDARY OUTCOMES:
Neurologic outcomes at hospital discharge | upto 24 weeks
  Patient who suffered in hospital cardiac arrest has variable neurologic outcomes. This will be evaluated with Glasgow outcome scale (GOS). This score ranges from 1 to 5 where GOS 1-3 is considered unfavourable neurologic outcomes and GOS 4-5 are considered favourable neurologic outcomes.
short term survival | upto 24 weeks
  Short term survival will include survival from hospital to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jignesh K Patel, MD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, South Setauket, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patel JK, Schoenfeld E, Hou W, Singer A, Rakowski E, Ahmad S, Patel R, Parikh PB, Smaldone G. Inhaled nitric oxide in adults with in-hospital cardiac arrest: A feasibility study. Nitric Oxide. 2021 Oct 1;115:30-33. doi: 10.1016/j.niox.2021.07.001. Epub 2021 Jul 3. PMID 34229057
- [Derived] Magliocca A, Fries M. Inhaled gases as novel neuroprotective therapies in the postcardiac arrest period. Curr Opin Crit Care. 2021 Jun 1;27(3):255-260. doi: 10.1097/MCC.0000000000000820. PMID 33769417